CLINICAL TRIAL: NCT04542642
Title: A Randomized, Controlled, Open-Label, Decentralized Study, to Evaluate Patient Engagement With PEAR-008, a Game-Based Digital Therapeutic for the Treatment of Opioid Use Disorder
Brief Title: A Remote, Decentralized Opioid Use Disorder Study to Evaluate Patient Engagement With a Game-Based Digital Therapeutic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pear Therapeutics, Inc. (Industry)
Collaborators: Addiction Research and Education Foundation (AREF) (Unknown); Research Foundation for Mental Hygiene, Inc. (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PEAR-008-101; R44DA042652 (NIH)
Record Dates: First submitted 2020-08-27; First posted 2020-09-09 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Opioid-use Disorder
Keywords: digital therapeutic
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to receive either the game-based treatment (PEAR-008) or the original, FDA-authorized treatment (reSET-O).
Who Masked: Outcomes Assessor
Masking Description: Independent Outcomes Assessor will conduct data analysis and be blinded to intervention assignments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- reSET-O (Active Comparator): Prescription Digital therapeutic
  Interventions: Device: reSET-O
- PEAR-008 (Experimental): Investigational Digital Therapeutic
  Interventions: Device: PEAR-008

INTERVENTIONS:
Device: reSET-O — reSET-O is an FDA-authorized mobile application treatment for opioid use disorder.
  Arms: reSET-O
Device: PEAR-008 — PEAR-008 is a new, game-based version of reSET-O, a mobile application treatment for opioid use disorder.
  Arms: PEAR-008

SUMMARY:
The purpose of this study is to evaluate how patients use and engage with a game-based mobile application that is designed to treat opioid use disorder.

DETAILED DESCRIPTION:
This is a randomized, controlled, open-label, decentralized study to evaluate patient engagement with PEAR-008, a game-based digital therapeutic for the treatment of opioid use disorder.

PEAR-008 is a new version of reSET-O, an FDA-authorized mobile application treatment (available by prescription only) for opioid use disorder. The study will examine if changing the application's delivery format and enhancing clinical content affects how patients use and interact with the intervention.

Prospective participants will complete a short screening assessment and if eligible complete informed consent procedures at the beginning of the Baseline visit. Qualifying participants will attend weekly virtual study visits during the 8-week treatment period.

In addition to weekly assessments, additional assessments will be administered at week 4 and week 8. Participants will be asked to complete a follow-up assessment 4 weeks after completing treatment.

ELIGIBILITY:
Inclusion Criteria:

* Provide informed consent prior to any study specific assessments being performed
* Between 18 and 60 years old, inclusively
* Proficient in English language
* Within the first 120 days of starting buprenorphine treatment
* Receiving buprenorphine pharmacotherapy under the care of a licensed healthcare provider and willing to provide the provider or practice name
* Capable of using common software applications on a mobile device (smartphone)
* Access to an internet-enabled smartphone for the duration of the study, meeting minimal operations systems (OS) requirements
* Interest in using a digital therapeutic for Opioid-use Disorder
* No prior history of reSET-O use
* Has not participated in user testing of PEAR-008 or any investigational drug trials within the past 30 days of enrollment

Exclusion Criteria:

* On methadone or naltrexone pharmacotherapy
* Unable to use English to participate in the consent process, interventions, or assessments
* Inability to comply with study procedures

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2021-05-19 (Actual); Primary Completion 2022-11-16 (Actual); Study Completion 2022-11-23 (Actual)

PRIMARY OUTCOMES:
Evaluate Participant Engagement Data | From Week 1 to Week 8 (End of Treatment)
  Evaluate the number of active sessions per week between PEAR-008 and reSET-O

SECONDARY OUTCOMES:
Evaluate Treatment Retention Based on Drop-Out Rates | Week 1, Week 2, Week 3, Week 4, Week 5, Week 6, Week 7, Week 8 (End of Treatment), Week 12 (Follow-up)
  Evaluate if PEAR-008 increases retention in treatment compared to reSET-O by comparing drop-out rates
Evaluate Illicit Drug Abstinence | Week 1, Week 2, Week 3, Week 4, Week 5, Week 6, Week 7, Week 8 (End of Treatment), Week 12 (Follow-up)
  Evaluate if PEAR-008 increases abstinence compared to reSET-O, as measured by saliva drug screens, urine drug screens and self-reporting
Evaluate Digital Therapeutic Use Patterns Based on Usage Data | From Week 1 to Week 8 (End of Treatment)
  Evaluate participants' digital therapeutic use patterns based on usage data collected, comparing PEAR-008 to reSET-O
Assess Effect on Depressive Symptoms | Baseline, Week 4, Week 8 (End of Treatment), Week 12 (Follow-up)
  Assess the effect of PEAR-008 and reSET-O on depressive symptoms using the eight-item Patient Health Questionnaire (PHQ-8) scores from Baseline to End of Treatment and Follow-up. The PHQ's total score ranges from 0 (not clinically significant) to 24 (clinically significant)
Assess Effect on Anxiety Symptoms | Baseline, Week 4, Week 8 (End of Treatment), Week 12 (Follow-up)
  Assess the effect of PEAR-008 and reSET-O on anxiety symptoms using the Generalized Anxiety Disorder-7's (GAD-7) scores from Baseline to End of Treatment and Follow-up. The GAD-7's total score ranges from 0 (not clinically significant) to 21 (clinically significant)
Assess Effect on Recovery Capital | Baseline, Week 4, Week 8 (End of Treatment), Week 12 (Follow-up)
  Assess the effect of PEAR-008 and reSET-O on recovery capital using the ten-item Brief Assessment of Recovery Capital (BARC-10) scores from Baseline to End of Treatment and Follow-up. The BARC-10's total score ranges from 10 to 60
Describe Participant Satisfaction Surveys | Baseline, Week 4, Week 8 (End of Treatment), Week 12 (Follow-up)
  Summarize participant satisfaction surveys and evaluate if PEAR-008 increases participant satisfaction in treatment compared to reSET-O through descriptive statistics
Describe Participant Satisfaction Interviews | Week 12 (Follow-up)
  Summarize participant satisfaction interviews and evaluate if PEAR-008 increases participant satisfaction in treatment compared to reSET-O through descriptive statistics
Assess Coronavirus Disease (COVID-19) Impact | Baseline, Week 4, Week 8 (End of Treatment), Week 12 (Follow-up)
  Assess the impact of the COVID-19 pandemic on participants using the five-item Council on American-Islamic Relations (CAIR) Pandemic Impact Questionnaire (C-PIQ) scores from Baseline to End of Treatment and Follow-up. The C-PIQ's total score ranges from 0 to 20
Assess Coronavirus Disease (COVID-19) Impact on Stress | Baseline, Week 4, Week 8 (End of Treatment), Week 12 (Follow-up)
  Assess the effect of the COVID-19 pandemic on depressive symptoms using the COPE: Coronavirus Perinatal Experiences - Impact Survey (COPE-IS) (MODIFIED) scores from Baseline to End of Treatment and Follow-up. Participants will be asked how they are coping with stress during COVID-19 from a list of responses. There is no scoring for this measure
Assess Effect on Resilience | Baseline, Week 4, Week 8 (End of Treatment), Week 12 (Follow-up)
  Assess the effect of PEAR-008 and reSET-O on resilience using the 10-item Connor-Davidson Resilience Scale 10 (CD-RISC-10) scores from Baseline to End of Treatment and Follow-up. The CD-RISC-10 is a 10-item self-rating scale using a 5-point Likert scale ranging from "not true at all" to "true nearly all of the time"

OTHER OUTCOMES:
Evaluate Engagement and Efficacy Relationship | From Week 1 to Week 8 (End of Treatment), Week 12 (Follow-up)
  Evaluate the correlation between engagement (daily and weekly participant use patterns of PEAR-008 and reSET-O) and treatment outcomes (abstinence and retention in treatment)
Change in Skill Acquisition | Baseline, Week 4, Week 8 (End of Treatment), Week 12 (Follow-up)
  Assess the effect of PEAR-008 and reSET-O on changes in skill acquisition using the Cognitive-Behavioral Therapy Skills Questionnaire (CBTSQ) from Baseline to End of Treatment. The CBTSQ measures two factors: Behavioral Activation (BA) and Cognitive Restructuring (CR). BA factor scores range from 0 to 35, and higher scores indicate greater use of BA skills. CR factor scores range from 0 to 45, and higher scores indicate greater use of CR skills
Medication Adherence Rates | Week 1, Week 2, Week 3, Week 4, Week 5, Week 6, Week 7, Week 8 (End of Treatment), Week 12 (Follow-up)
  Assess the effect of PEAR-008 and reSET-O on medication adherence rates using findings from saliva drug screens and urine drug screens

CONTACTS AND LOCATIONS:
Overall Officials: Aimee Campbell, PhD, Study Director — Columbia University; Lisa Chiodo, PhD, Study Director — Addiction Research and Education Foundation
Locations (2):
- United States (2):
  - The Substance and Treatment Research Service (STARS) at Columbia University Irving Medical Center and the New York State Psychiatric Institute, New York, New York
  - Addiction Research and Education Foundation, Gig Harbor, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Luderer H, Chiodo L, Wilson A, Brezing C, Martinez S, Xiong X, Gerwien R, Imbert B, Deeg M, Maricich Y, Campbell A. Patient Engagement With a Game-Based Digital Therapeutic for the Treatment of Opioid Use Disorder: Protocol for a Randomized Controlled Open-Label, Decentralized Trial. JMIR Res Protoc. 2022 Jan 26;11(1):e32759. doi: 10.2196/32759. PMID 35080499